CLINICAL TRIAL: NCT06904066
Title: A Phase I Study of Autologous T Cells Transduced With Retroviral Vectors Expressing TCRs for Participant-specific Neoantigens in Patients With Acute Myeloid Leukemia, Myelodysplastic Syndrome, and Other Hematologic Malignancies
Brief Title: Autologous T Cells Transduced With Retroviral Vectors Expressing TCRs for Participant-specific Neoantigens in Patients With Hematologic Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10002088; 002088-C
Record Dates: First submitted 2025-03-29; First posted 2025-04-01 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-20

CONDITIONS: Malignancy, Hematologic; Neoplasms, Hematologic; Neoplasms, Hematopoietic; Blood Cancer; Hematological Neoplasms; Hematopoietic Malignancies; Dysmyelopoietic Syndromes; Hematopoetic Myelodysplasia; Myeloid Leukemia, Acute; Nonlymphoblastic Leukemia, Acute; Leukemia, Lymphocytic, Acute
Keywords: Gene Therapy; T cell immunotherapy; Engineered T cell receptor; Hematologic Malignancies; Tumor-Associated Antigen; Myelodysplastic Syndrome; Neoepitope-specific T cells; T-cell acute lymphoblastic leukemia; Adoptive T Cell Therapy; Chronic Myeloid Leukemia
MeSH Terms: conditions — Hematologic Neoplasms; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — aldesleukin; Cyclophosphamide; fludarabine phosphate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- 1/Experimental: No allo-HSCT (Experimental): Preparative regimen of cyclophosphamide and fludarabine + infusion of neoepitope-specific T cells (of up to 1.5x10^11 total cells) + aldesleukin.
  Interventions: Drug: aldesleukin; Drug: cyclophosphamide; Drug: fludarabine phosphate; Biological: Individual Patient TCR-Transduced PBL; Device: TruSight Oncology (TSO) 500
- 2/Experimental: prior allo-HSCT (Experimental): Preparative regimen of cyclophosphamide and fludarabine + infusion of neoepitope-specific T cells (at a dose of 1x10^10 total cells) + aldesleukin.
  Interventions: Drug: aldesleukin; Drug: cyclophosphamide; Drug: fludarabine phosphate; Biological: Individual Patient TCR-Transduced PBL; Device: TruSight Oncology (TSO) 500

INTERVENTIONS:
Drug: aldesleukin — Aldesleukin 600,000 IU/kg IV (based on total body weight) over 15 minutes approximately every 8 hours beginning within 24 hours of cell infusion and continuing for up to 4 days (maximum 10 doses).
Drug: cyclophosphamide — 300 mg/m^2 IV infusion over 30 minutes. Daily x 3 doses on days -5, -4, -3.
Drug: fludarabine phosphate — 30 mg/m^2 IV infusion over 30 minutes administered immediately following cyclophosphamide on day -5, -4, -3. Participants with renal dysfunction receive a lower dose of fludarabine.
Biological: Individual Patient TCR-Transduced PBL — Up to 1.5x10^11 total cells for non-transplant subjects. 1x10^10 total cells for post-alloHSCT subjects.
Device: TruSight Oncology (TSO) 500 — TSO500 sequencing panel performed in the NCI Laboratory of Pathology to detect TP53 or RAS mutations

SUMMARY:
Background:

Blood cancers (such as leukemias) can be hard to treat, especially if they have mutations in the TP53 or RAS genes. These mutations can cause the cancer cells to create substances called neoepitopes. Researchers want to test a method of treating blood cancers by altering a person s T cells (a type of immune cell) to target neoepitopes.

Objective:

To test the use of neoepitope-specific T cells in people with blood cancers

Eligibility:

People aged 18 to 75 years with any of 9 blood cancers.

Design:

Participants will have a bone marrow biopsy: A sample of soft tissue will be removed from inside a pelvic bone. This is needed to confirm their diagnosis and the TP53 and RAS mutations in their cancer cells. They will also have a skin biopsy to look for these mutations in other tissue.

Participants will undergo apheresis: Blood will be taken from their body through a vein. The blood will pass through a machine that separates out the T cells. The remaining blood will be returned to the body through a different vein.

The T cells will be grown to become neoepitope-specific T cells.

Participants receive drugs for 3 days to prepare their body for the treatment. The modified T cells will be given through a tube inserted into a vein. Participants will need to remain in the clinic at least 7 days after treatment.

Participants will have 8 follow-up visits in the first year after treatment. They will have 6 more visits over the next 4 years. Long-term follow-up will go on for 10 more years.

DETAILED DESCRIPTION:
Background:

* Many difficult-to-treat hematologic malignancies carry mutations in the tumor suppressor gene TP53 or the oncogenes NRAS and KRAS (shortened to RAS).
* Missense mutations in TP53 and RAS result in immunogenic peptides (neoepitopes) that can be presented by human leukocyte antigens (HLA) to initiate an immune response.
* The NCI Surgery Branch has previously identified T-cell receptors (TCRs) that selectively recognize p53 or Ras neoepitopes.
* We propose to evaluate 3 TCRs targeting p53 neoepitopes and 4 TCRs targeting Ras neoepitopes in participants with hematologic malignancies.
* Several of these TCRs have already been evaluated in clinical trials enrolling subjects with solid tumors.
* We have shown that the TCRs have activity against hematologic malignancy cell lines in vitro and in vivo and have high specificity for only cells expressing the targeted mutation and the correct HLA.

Primary Objective:

-To determine the safety of administering neoepitope-specific T cells targeting p53 or Ras neoepitopes in combination with preparative conditioning chemotherapy and aldesleukin in participants with hematologic malignancies

Eligibility:

Participants must be/have:

* Myelodysplastic syndrome, acute myeloid leukemia, chronic myeloid leukemia, chronic myelomonocytic leukemia, T-cell acute lymphoblastic leukemia/lymphoma, or multiple myeloma
* Age >=18 and <=75 years old
* The malignant cells must have a mutation in TP53 or RAS at a location targeted by one of a panel of TCRs.
* The participant must have the HLA type capable of presenting the targeted neoepitope.
* Recipients with relapsed or persistent malignancy after previous HLA-matched sibling or matched unrelated donor allogeneic hematopoietic stem cell transplant (alloHSCT) are eligible.
* AlloHSCT recipients must not have evidence of acute graft-versus-host disease (GVHD).
* AlloHSCT recipients must have no chronic GVHD or mild chronic GVHD as defined by NIH Consensus Development Project Criteria.
* Circulating malignant cells (blasts or plasma cells) must be 1% or less of peripheral white blood cells.

Design:

* This is an open-label, single center, non-randomized phase I trial
* Peripheral blood mononuclear cells (PBMCs) will be harvested by leukapheresis and cultured with anti-CD3 (OKT3) and aldesleukin to stimulate T-cell growth.
* The T cells will be genetically modified using a replication-incompetent gamma-retrovirus encoding a TCR.
* All participants will receive a chemotherapy conditioning regimen of cyclophosphamide and fludarabine.
* After the chemotherapy ends, participants will receive an infusion of the neoepitope-specific T cells and begin aldesleukin infusions.
* Following neoepitope-specific T-cell infusion, there is a mandatory inpatient hospitalization to monitor for toxicity.
* Frequent outpatient follow-up and malignancy assessment is planned after treatment.

ELIGIBILITY:
* INCLUSION CRITERIA:

Malignancy diagnosis requirements:

-Eligible diagnoses include AML (acute myeloid leukemia), MDS (myelodysplastic syndrome), CMML(chronic myelomonocytic leukemia), CML (chronic myeloid leukemia), and T-ALL (T-acute lymphoblastic leukemia/lymphoma) meeting standard diagnostic criteria as described in the 5th edition World Health Organization Classification of Hematologic Tumors and/or the International Consensus Classification of Myeloid Neoplasms and Acute Leukemias. Multiple myeloma participants meeting International Working Group diagnostic criteria are eligible. These diagnostic criteria can be met at any time during the course of the participant s malignancy. Atypical CML is not an eligible diagnosis.

NOTE: Pathology reports are acceptable to confirm eligibility.

Malignancy mutation and HLA requirements:

* Detection of at least one of the neoepitope-forming TP53 or RAS mutations that are listed in Table 3 in on the TruSight Oncology (TSO) 500 sequencing panel (NSR device) performed in the NCI Laboratory of Pathology is required. RAS mutations can be in NRAS, KRAS or HRAS as these oncogenes have the same amino acid sequence at the location of the targeted neoepitopes. A variant allele frequency (VAF) of at least 5% is required for a mutation to be eligible. This criterion can be met at any time within 60 days prior to apheresis regardless of treatment history during this 60-day period. DNA for sequencing comes from bone marrow.
* Presence of the correct HLA type needed to present one of the targeted neoepitopes as shown in Table 3. HLA typing data from any time-point prior to apheresis can be used to meet this requirement.

Table 3: Eligibility requirements for the targeted mutation and HLA type

Targeted mutation - TP53 R175H; HLA Type - A*02:01

Targeted mutation - TP53 Y220C; HLA Type - A*02:01

Targeted mutation - TP53 R248W; HLA Type - A*68:01

Targeted mutation - Ras G12V; HLA Type - A*11:01

Targeted mutation - Ras G12D; HLA Type - A*11:01

Targeted mutation - Ras G12D; HLA Type - C*08:02

Targeted mutation - Ras G12V; HLA Type - C*01:02

Malignancy burden requirements:

* For AML and MDS, bone marrow myeloblast percentage must be >=5% of nucleated cells in either bone marrow aspirate or biopsy. Myeloblasts can be defined by immunohistochemistry or by cytochemistry stains including but not limited to myeloperoxidase.
* For T-ALL, bone marrow T-cell blast percentage must be >=5% of nucleated cells in either bone marrow aspirate or biopsy. T cells can be defined by cytochemistry or immunohistochemistry or flow cytometry.
* For multiple myeloma, plasma cells having a phenotype consistent with multiple myeloma must be detected at any frequency by multiparameter bone marrow flow cytometry or total plasma cells must be at least 6% on bone marrow core biopsy or bone marrow aspirate.
* For CMML, bone marrow blast (including monocytic blast equivalent) percentage must be >=6% of bone marrow nucleated cells by cytochemistry or immunohistochemistry of bone marrow aspirate or biopsy.
* For CML measurable leukemia is defined as molecular detection of BCR-ABL1 at a ratio of >1.0% to ABL1 or another housekeeping gene on The International Scale (IS) in either blood or bone marrow.

Malignancy prior treatment and risk category criteria

- Participants with AML, MDS, CML, CMML, and T-ALL who have not had prior allogeneic hematopoietic stem cell transplantation (alloHSCT) must be unwilling or unable to undergo alloHSCT.

NOTE: Unable to undergo alloHSCT could be due to lack of access to transplantation or not meeting transplant eligibility criteria at one or more transplant centers where the participant was evaluated by a transplant physician.

* Participants with primary, secondary, or treatment-related AML that did not go into remission after induction therapy are eligible regardless of history of alloHSCT.
* Myelodysplastic syndrome (MDS)

  * Participants with MDS must have had high or very high risk MDS as determined by IPSS-R or IPSS-M (https://mds-risk-model.com) at any time point.
  * Participants with MDS must have received previous treatment with at least one of the following: a hypomethylating agent, cytotoxic chemotherapy, or alloHSCT. Participants with primary or treatment-related MDS are eligible.
  * Participants with MDS/AML with mutated TP53 are eligible.
* Participants with CMML must have had a CMML-specific prognostic scoring system-Molecular (CPSS-Mol) score of >=2 (Intermediate-2 or High risk groups) at any time-point and must have received at least one line of previous systemic treatment, which could have been alloHSCT.
* Chronic myeloid leukemia (CML)

  * Participants with chronic phase CML and a history of inadequate response to or intolerance of 3 or more tyrosine kinase inhibitors (TKIs) are eligible.
  * In addition, participants who have received at least one of bosutinib, dasatinib, or nilotinib in addition to either ponatinib or asciminib are eligible. Participants in accelerated phase or blast crisis are eligible if they have received at least one TKI.
  * Participants who have received a prior HSCT are eligible provided they have also received at least 2 TKIs and meet other eligibility criteria.
* Participants with T-ALL must have T-ALL that did not go into CR with induction therapy or that relapsed.
* Participants with relapsed AML who are unable to undergo alloHSCT and meet other eligibility requirements are eligible.
* Multiple Myeloma

  * Participants with multiple myeloma must have received at least 3 different prior systemic treatment regimens for multiple myeloma. Participants must have prior exposure to an imid such as lenalidomide, a proteosome inhibitor, and a BCMA-targeting CAR T-cell therapy, such as monoclonal antibody, or bispecific antibody.
  * Multiple myeloma participants with a history of alloHSCT are eligible
  * Participants with multiple myeloma must also have measurable multiple myeloma

defined by at least one of the criteria below:

* Serum M-protein greater or equal to 1.0 g/dL.
* Urine M-protein greater or equal to 200 mg/24 h.
* Serum free light chain (FLC) assay: involved FLC level greater or equal to 10mg/dL (100 mg/L) provided serum FLC ratio is abnormal.
* A biopsy-proven plasmacytoma at least 2.0 cm in largest dimension.
* Bone marrow core biopsy with 30% or more plasma cells.

Other inclusion criteria

* Blast cells <=1% of white blood cells as measured by CBC and differential before apheresis
* Plasma cells <=1% of white blood cells as measured by CBC and differential before apheresis
* Participants must be willing to undergo intensive care unit care including mechanical ventilation if necessary
* Participants must not have received systemic chemotherapy for at least 14 days prior to start of lymphodepleting chemotherapy or apheresis, and chemotherapy-related toxicities other than cytopenias must have recovered to grade 0 or grade 1 by the time of apheresis. The one exception is if necessary to control AML, CML, or CMML, hydroxyurea can be administered up to 7 days prior to apheresis.
* Participants who have received alloHSCT must have received a transplant from either a fully matched sibling or 10/10 HLA-matched unrelated donor.
* Recipients of alloHSCT must be at least 100 days post-transplant before the apheresis.
* Subjects must be willing to be co-enrolled on NCI protocol 03C0277 and 09C0161.
* Age must be >=18 and <= 75 years old
* Clinical performance status of ECOG 0 or 1
* Participants must have adequate organ function as defined below:

  * Hemoglobin: >=8 g/dL without red blood cell transfusions for 7 days prior to blood count check
  * Platelets: >=45,000/mcL without transfusion support in the 7 days prior to the blood count check
  * Absolute neutrophil count: >=850/mcL without exogenous growth factor administration within the 10 days prior to the blood count check
  * Total bilirubin: <= 2.0 mg/dL. Except for participants with Gilbert s syndrome (who must have a total bilirubin <3 mg/dL)
  * Alanine transaminase (ALT) and aspartate transaminase (AST): <= to 3 times the upper limit of the institutional normal unless liver involvement by malignancy is demonstrated. If liver involvement with malignancy is detected, ALT and AST must be <= 5 times the upper limit of normal
  * Serum Creatinine: <= 1.5 mg/dL
* Participants who have received prior genetically-engineered T-cell therapies are eligible if at least 180 days have elapsed between the date of previous T-cell infusion and apheresis.
* Room air oxygen saturation must be 93% or greater
* Women of child-bearing potential (WOCBP) must agree to use highly effective contraception (hormonal, intrauterine device [IUD], abstinence, surgical sterilization) starting at the time of study entry, for the duration of study therapy, and 12 months after the last dose of combined chemotherapy. NOTE: IOCBP is defined as any person who has experienced menarche and who has not undergone successful surgical sterilization or who is not postmenopausal.

Men able to father children must agree to use an effective method of contraception (barrier, surgical sterilization, abstinence) for the duration of the study treatment and for 4 months after the last dose of combined chemotherapy. We also will recommend these Men with partners of childbearing potential ask their partners to be on highly effective birth control (hormonal, intrauterine device [IUD], surgical sterilization). Men able to father a child must not freeze or donate sperm within the same period.

* Nursing participants must be willing to discontinue breastfeeding from study treatment initiation through 4 months after the last dose of the study drug(s).
* Hepatitis B surface antigen and hepatitis B core antibody tests must be negative. If either of these tests are positive, participants must have a negative blood PCR test for hepatitis B to enroll on the study.
* Hepatitis C antibody test must be negative. If this test is positive, participants must have a negative blood PCR test for hepatitis C RNA to enroll on the study.
* Cardiac ejection fraction of greater than or equal to 50% by echocardiography with no evidence of hemodynamically significant pericardial effusion as determined by an echocardiogram within 30 days prior to apheresis.
* All participants must be willing to undergo mandatory bone marrow biopsy/ aspirates during the study.
* Participants with a history of cigarette smoking of >5 pack years, a history of pulmonary disease, a history of alloHSCT, or chronic pulmonary symptoms must undergo pulmonary function testing and have an FEV1 >50% predicted and diffusing capacity for carbon monoxide >= 60%.
* Subjects who received a previous allogeneic HSCT must have no (grade 0) acute GVHD and no chronic GVHD or mild chronic GVHD as defined.

  --NOTE: Subjects with GVHD meeting the above criteria with local therapy (topical cutaneous steroids, inhaled steroids, and eye drops) will be eligible.
* Potential participants must agree to stay within 1-hour drive of NIH clinical center from date of initial discharge until at least 14 days have elapsed since T cell infusion through the 14 day time period.
* Ability of the participant to understand and the willingness to sign a written informed consent document.
* Willing to sign a durable power of attorney.

EXCLUSION CRITERIA:

-For alloHSCT recipients only, subjects receiving any systemic immunosuppressive drugs including corticosteroids at doses of greater than 5 mg/day prednisone or equivalent within 28 days prior to apheresis.

NOTE: Topical corticosteroid preparations applied to the skin such as solutions, creams, and ointments are allowed. Inhaled corticosteroids are allowed, and corticosteroid eye drops are allowed.

* Corticosteroids given for any indication at doses greater than 5 mg/day of prednisone or equivalent within 14 days before either apheresis or start of protocol chemotherapy.
* Participants with MDS/Myeloproliferative neoplasia overlap syndromes are not eligible.
* Participants with acute promyelocytic leukemia are not eligible.
* Participants who received a mis-matched sibling or haploidentical transplant are not eligible.
* Tumor masses >=10 cm in largest diameter
* Positive beta Human chorionic gonadotropin (beta-HCG) serum or urine pregnancy test in IOCBP performed at screening.
* Human T-cell lymphotropic virus type 1/ 2 (HTLV-1/II) positive
* HIV infection, as measured by seropositivity for HIV antibody.
* Participants that require urgent therapy due to tumor mass effects on vital organ or tumor lysis syndrome.
* Any significant illness that, in the opinion of the principal investigator, may impair the participant s tolerance of the study treatment as evaluated by medical history, physical exam, assess for hepatosplenomegaly, and chemistry laboratory evaluations.
* Participants with a history of a previous malignancy are ineligible if the malignancy has not been in complete remission for at least 2 years or if the previous malignancy required treatment with surgery, radiation, or chemotherapy, including maintenance hormonal therapy, in the past 2 years. Exceptions to this requirement are participants who have had successful resection of the following types of skin cancer: nonmetastatic basal cell carcinoma or squamous cell carcinoma or stage 0 melanoma.
* Suspected or confirmed active uncontrolled infections defined as fevers of >38 degrees within the past 24 hours without a known non-infectious source or participants requiring intravenous antibiotics when intravenous antibiotics have been administered for less than 72 hours.
* Acti...

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Safety | From time of the lymphodepleting chemotherapy through 5 years after neoepitope-specific T cell infusion or until off study.
  Adverse Events (AE) per CTCAE v5.0, by type, grade, and frequency

SECONDARY OUTCOMES:
Overall response rate | up to 5 years
  Defined by the Overall Response Rate (CR+PR) and the CR rate, duration of response. Duration of response will be calculated from the first date of a response until relapse, progression, or initiation of a new anti-malignancy therapy
Feasibility of manufacturing and administering neoepitope-specific T cells | 30 days post treatment completion
  Feasibility will be measured as the fraction of participants with successful infusion of neoepitope-specific T-cell. Successful neoepitope-specific T-cell infusion will be achieved when at least 1x10^10 total cells are infused

CONTACTS AND LOCATIONS:
Overall Officials: James N Kochenderfer, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the NIH Data Management and Sharing (DMS) Policy, which applies to all new and ongoing NIH-funded research in the IRP, as of January 25, 2023, that is associated with a ZIA, with a clinical protocol that undergoes scientific review and/or will involve genomic data sharing. @@@@@@@@@@@@This study will comply with the NIH Genomic Data Sharing (GDS) Policy, which applies to all new and ongoing NIH IRP-funded research, as of January 25, 2015, that generates large-scale human or non-human genomic data, as well as the use of these data for subsequent research. Large-scale data include genome-wide association studies (GWAS), single nucleotide polymorphisms (SNP) arrays, and genome sequence, transcriptomic, epigenomic, and gene expression data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be available until completion of the primary endpoint.
Access Criteria: Clinical data will be made available with the permission of the study PI. Clinical data at NIH will also be available via subscription to BTRIS.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_002088-C.html